CLINICAL TRIAL: NCT04303637
Title: The Impact of Phone Use on Everyday Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yale-NUS College (Other)
Responsible Party: Principal Investigator, Jean Liu, Assistant Professor, Yale-NUS College
Other Study IDs: S-18-213
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Sleep; Depression; Anxiety
Keywords: Smartphone; Screen time
MeSH Terms: conditions — Obesity; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High school student: 13-18 year old students enrolled in schools within Singapore.
  Interventions: Behavioral: Phone use

INTERVENTIONS:
Behavioral: Phone use — Objective and subjective reports of smartphone use (e.g., number of hours, number of pick-ups, how phones are used)

SUMMARY:
Participants will download a phone-tracking app for a week to track phone usage, providing objective data on usage patterns. Quantitative tasks and questionnaires will also be carried out before and after the tracking period.

DETAILED DESCRIPTION:
A notable shortcoming of existing mobile phone research is that 'phone use' has almost exclusively been measured through subjective reports - by simply asking respondents how much time they spend on their mobile phones each day. This operational definition, however, is a major shortcoming as phone use is difficult to track - and is thus likely to be highly inaccurate.

To address this gap, the investigators describe in this proposal a first step to characterize phone usage in an objective manner - by asking adolescents to download a phone-tracking app for a week. This circumvents measurement errors inherent to self-reports, and allows us to probe: (1) how accurate adolescents' estimates are of their own phone usage, and (2) whether objective phone usage predicts any cognitive, socio-emotional, or physical outcomes. The completion of this study will represent an important step forward in the development of empirically-driven guidelines on phone use amongst adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Owns a smartphone

Exclusion Criteria:

* Parents not willing to give consent
* History of medical or psychiatric disorder
* History of motion sickness, dizziness or epilepsy

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents aged 13-18 years old recruited from Singapore schools.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-06-10 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale (DASS 21) | 11 minutes (single measurement)
  A 21-item, 4-point scale measuring participant emotional states. This is the short form of the longer 42-item DASS.
Body mass index | 1 minute (single measurement)
  Participants' body mass index
Sleep duration | 2 minute (single measurement)
  Assessment of participants' sleep time & wake time

SECONDARY OUTCOMES:
Digit Span Task | 10 minutes (single measurement)
  A digit span task carried out using a computer program
Psychomotor Vigilance Task | 10 minutes (single measurement)
  PVT carried out using a computer program
Pediatric Daytime Sleepiness Scale (PDSS) | 5 minutes (single measurement)
  A 8-item, 5-point self-report scale to measure sleepiness during the day.
Strengths and Difficulties Questionnaire (SDQ) | 10 minutes (single measurement)
  A questionnaire looking at a student's emotional and behavioural aspects in relation to coping with school.

OTHER OUTCOMES:
General Questionnaire on Media Consumption | 5 minutes (single measurement)
  A short questionnaire on the usage patterns of various media devices.
Subjective Report of Phone Usage | 10 minutes (single measurement)
  A 5-item questionnaire that collects data on self-reported phone use patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Liu, PhD, Principal Investigator — Yale-NUS College
Locations (1):
- Yale-NUS College, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Stipulations by the institutional review board do not allow individualized data to be shared.